CLINICAL TRIAL: NCT07247604
Title: Pattern of Congenital Heart Diseases and Developmental Evaluation in Children Below Two Years With Cholestasis at Assiut University Children's Hospital
Brief Title: Congenital Heart Diseases and Developmental Assessment in Cholestatic Infants Under Two Years
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ahmed Mahros, Resident, Family Medicine Department, Assiut University
Other Study IDs: CHD-CHOLEST-ASSIUT
Record Dates: First submitted 2025-11-15; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cholestasis; Congenital Heart Disease
MeSH Terms: conditions — Cholestasis; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart diseases (CHDs) are common in infants with cholestasis due to shared prenatal and metabolic factors. This study aims to determine the frequency and types of CHDs and to assess physical and mental development in children below two years with cholestasis at Assiut University Children's Hospital.

DETAILED DESCRIPTION:
Congenital heart diseases (CHDs) are the most common structural malformations in childhood, affecting approximately 8-12 per 1,000 live births worldwide. Infants with systemic disorders such as neonatal and infantile cholestasis have a higher prevalence of CHDs due to overlapping prenatal insults, genetic syndromes, and metabolic disturbances. Cholestasis, defined as impaired bile flow with conjugated hyperbilirubinemia, may arise from biliary atresia, neonatal hepatitis, or metabolic and syndromic disorders such as Alagille syndrome. Several studies highlight a strong association between cholestasis and CHDs, and early recognition of this dual burden is essential to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children below 2 years presenting with cholestasis

Exclusion Criteria:

* Prematurely born infants.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with various causes of cholestatic disorders evaluated for congenital heart diseases and developmental outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Frequency of CHDs among cholestatic infants | At initial clinical evaluation
  Assessment of prevalence of congenital heart diseases in infants below 2 years with cholestasis.

SECONDARY OUTCOMES:
Types of CHDs identified in cholestatic infants | During hospital evaluation
  At baseline echocardiographic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mahran Mohammed, Prof., Study Chair — Professor of Family Medicine

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive clinical information about pediatric patients, and sharing is not permitted by the institutional ethics committee.